CLINICAL TRIAL: NCT01462682
Title: Perception of Fatigue Among Surgeons During Night Shifts, a Focus Group Study.
Brief Title: Perception of Fatigue Among Surgeons During Night Shifts
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Principal Investigator, Ilda Amirian, MD, PHD student at Unit of Surgical Gastroenterology, Herlev Hospital
Other Study IDs: Herlev-1234
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2011-12

CONDITIONS: Fatigue
Keywords: focus group study; sleep deprivation; surgery
MeSH Terms: conditions — Fatigue; Sleep Deprivation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to illustrate surgeons' own perception of fatigue and the impact they felt it had on their performance. This was accomplished through a focus group study, where 13 surgeons participated.

ELIGIBILITY:
Inclusion Criteria:

* Doctors working at department of surgical gastrointerology, who gave informed consent

Exclusion Criteria:

* Withdrawal of consent

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Doctors working at a department of surgical gastroenterology
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Herlev Hospital, Herlev, Herlev, Denmark